CLINICAL TRIAL: NCT02162537
Title: Multicentric, Randomized, Phase III Trial Comparing 2 Strategies in Patients With Non-squamous Non-small Cell Lung Cancer With Asymptomatic Brain Metastases
Brief Title: Therapeutic Strategies in Patients With Non-squamous Non-small Cell Lung Cancer With Brain Metastases
Acronym: METAL2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow inclusions due in part to a change in practices. The first chemotherapy become a standard for patients with NSCL with asymptomatic brain metastases.
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Principal Investigator, Isabelle MONNET, Physician, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: METAL 2
Record Dates: First submitted 2014-03-21; First posted 2014-06-12 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer; Adenocarcinoma of Lung Metastatic to Brain; Cerebral Metastases
Keywords: Strategy; Radiotherapy; Chemotherapy; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (standard arm) (Other): Arm A: Initial Cerebral Radiotherapy and Chemotherapy (Cisplatin and pemetrexed with or without Bevacizumab)
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Bevacizumab; Radiation: Cerebral Radiotherapy
- Arm B (experimental arm) (Other): Arm B: Chemotherapy (Cisplatin and pemetrexed with or without Bevacizumab) and Cerebral Radiotherapy if clinical or radiological progression brain
  Interventions: Drug: Cisplatin; Drug: Pemetrexed; Drug: Bevacizumab; Radiation: Cerebral Radiotherapy

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 75 mg/m2 IV (with adequate hydration) on D1 every 3 weeks.
  Other Names: Cisplatine
Drug: Pemetrexed — 500mg/m² IV(10 min. infusion, preceded by the usual folic acid, vitamin B12 and corticosteroid premedication)on D1 every 3 weeks
  Other Names: Alimta
Drug: Bevacizumab — 7.5 mg/kg on D1 every 3 weeks. In case of eligibility for Bevacizumab, the latter will not be started until C2.
  Other Names: Avastin
Radiation: Cerebral Radiotherapy — Cerebral radiotherapy (encephalon in toto, 30 gy 10 sessions and 12 days) immediately after randomization before D1.If the number of brain metastases is less than or equal to 5 and less than or equal to 5 cm size, cerebral stereotactic radiotherapy condition may be proposed. The recommended interval between randomisation and D1 will be approximately 4 weeks.
  Other Names: Brain Radiotherapy

SUMMARY:
The patients carrying a complicated primary lung cancer brain metastases die in less than 3 months of delay disease in the absence of treatment. The median survival of these patients is approximately six months when the treatment associated with radiotherapy chemotherapy based on cisplatin is now the standard treatment. In most studies the patients die of their brain disease in one case only two, so it is likely that some patients do not require brain irradiation (prognosis in this case is linked to extra-cerebral disease ). The benefits for patients in group B (without systematic irradiation) are not to suffer the side effects of this radiation. The risks are in the same group to see brain metastases become symptomatic.

The role of cerebral radiotherapy in the patients treated with chemotherapy is unclear: should all patients be irradiated systematically (since the "reference" treatment is involved and with the aim of obtaining better control of the brain lesions and maintaining a better neurological status) or should only the patients showing cerebral progression be irradiated (avoidance of possibly useless brain radiotherapy and its side effects). The aim of this study is to better determine the position of cerebral radiotherapy in this context.

Main objective:

determine whether there is a difference in terms of progression-free survival between a therapeutic strategy with initial systematic brain radiotherapy followed by chemotherapy cis-platine/alimta + / - Bevacizumab and strategy with an initial chemotherapy cis-platine/alimta + / - Bevacizumab associated with brain radiotherapy only in cases of cerebral progression in patients with NSCLC with asymptomatic brain metastases

DETAILED DESCRIPTION:
This is a trial comparing two strategies with the aim to determine the best place for cerebral radiotherapy (initially or only systematic progression).

Arm A: Initial cerebral radiotherapy and chemotherapy, standard arm Arm B: Chemotherapy and Radiotherapy brain if clinical or radiological cerebral progression , experimental arm (The chemotherapy treatments are standard treatments using drugs with authorization in this indication)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically proven non-epidermoid, non-small cell lung cancer, non-EGFR (Epidermal Growth Factor Receptor)-mutated (or mutation test impracticable).
2. Patients with brain metastasis/metastases without neurosurgical indication.
3. Asymptomatic patients (without treatment or with stable steroids or antiepileptic treatments for ≥ 5 days prior to obtaining the baseline MRI of the brain, and ≥ 5 days prior to first dose of study treatment (Cycle 1, Day 1).
4. At least one lesion measurable according to the RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
5. ECOG (Eastern Cooperative Oncology Group) Performance Status 0 - 1
6. No previous chemotherapy for this cancer, apart from adjunctive chemotherapy more than 18 months ago.
7. Prior surgery is authorized in case of documented recurrence or progression.
8. Adequate biological functions (hematologic, platelets, hemoglobin, hepatic function, alkaline phosphatases, ASAT (Aspartate transaminase) and ALAT (Alanine Aminotransferase); creatinine clearance).
9. For women: Effective contraception for women of childbearing age during treatment and for 6 months following treatment.

   For men: They must be surgically sterile or accept the use of effective contraception until 6 months after the treatment period.
10. Patients of more than 18 years of age.
11. Estimated survival of at least 12 weeks.
12. Consent signed by the patient

Exclusion Criteria:

1. Patients presenting with a brain lesion eligible for curative treatment (neurosurgical).
2. Symptomatic brain metastasis/metastases in spite of symptomatic treatment.
3. Epidermoid carcinoma.
4. Con indication of Bevacizumab is furthermore
5. Patients presenting with a brain lesion eligible for curative treatment (neurosurgery or radiosurgery).
6. Symptomatic brain metastasis/metastases in spite of symptomatic treatment.
7. Epidermoid carcinoma.
8. Cons indication of Bevacizumab
9. Inability to take the folic acid or vitamin B12 vitamin supplementation or the dexamethasone premedication (or any equivalent corticosteroid), or any inability to comply with the study procedures.
10. History of cancer, with the exception of cervical cancer in situ, skin cancer other than melanoma, adequately treated low-grade prostatic cancer (Gleason score <6), unless this cancer was diagnosed and treated more than 5 years ago without any signs of recurrence.
11. Patients presenting with a systemic disorder which, in the investigator's opinion, compromises their participation in the study for reasons related to treatment safety or compliance.
12. Patients incapable of discontinuing their aspirin treatment when the dose is > 1300 mg/day or their non-steroidal anti-inflammatory treatment two days before the day, on the day and two days the day of administration of pemetrexed (Alimta).
13. Patients presenting with a 3rd sector (pleural effusion, ascites) which is clinically detectable and uncontrollable by simple measures of the evacuatory puncture type or other treatment before inclusion in the study.
14. Patients presenting with neuropathy of grade > 2 according to the criteria of CTC (Common toxicity Criteria) v3.0.
15. Patients whose foreseeable compliance or geographical distance renders monitoring difficult.
16. Pregnant or breast-feeding women.
17. Significant weight loss (≥ 10%) during the 6 weeks preceding inclusion in the study.
18. Vaccination against yellow fever within 30 days preceding inclusion in the study.
19. Cons-indication to taking steroids
20. Persons deprived of their liberty as a result of a judicial or administrative decision
21. Concomitant participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
To compare the progression-free survival rate in both arms | From date of the randomization until the date of first detection of progression, or until the date of death, assessed up to up to approximately 90 months
  Whether there is a difference in terms of progression-free survival between a therapeutic strategy with initial brain radiotherapy followed by systematic chemotherapy with cis-platinum / alimta and a strategy with initial chemotherapy with cis-platinum / alimta with brain radiotherapy only if brain progression in patients with non-small cell lung cancer with brain metastases asymptomatic.

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until the date of patient death, assessed up to 90 months
  After 4 cycles of chemotherapy with platinum salt-pemetrexed (with or without bevacizumab) possibly followed, in case of control of the disease and if the patient's condition allows, by pemetrexed (alone or with bevacizumab if the latter was part of the initial treatment) as maintenance treatment until progression.
Disease control rate (response + stability) | Baseline, between 21 and 28 days, then every 6 weeks, up to approximately 24 months
  Repeat examinations to assess the measurable lesions or initials and examination necessary to confirm the appearance of a new lesion in case of clinical suspicion of disease progression (minimum CT scan and MRI).The radiological treatment response will be measured according to the RECIST 1.1 criteria
Tolerance of treatment | Every 3 weeks, up to approximately 24 months
  The safety of the induction combination of cisplatin or carboplatin plus pemetrexed (Alimta®) +/- bevacizumab, the maintenance treatment with pemetrexed (Alimta®) +/- bevacizumab and the pancerebral radiotherapy will be assessed based on the CTC toxicity criteria v3.0.
Quality of life assessment | Baseline, between 21 and 28 days, then every 6 weeks, up to approximately 24 months
  The quality of life assessment measurement will be performed by self-questionnaire. The EURO-QOL questionnaire will be used.
Neurological assessment | Baseline, between 21 and 28 days, then every 6 weeks, up to approximately 24 months
  The neurological assessment measurement will be performed by self-questionnaire. The MOCA questionnaires will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle MONNET, Principal Investigator — Centre Hospitalier Intercommunal Créteil
Locations (41):
- France (41):
  - Centre Hospitalier, Charleville-Mézières, Ardennes
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre d'Oncologie et de Radiothérapie du Pays Basque, Bayonne
  - Centre Hospitalier, Beauvais
  - Hôpital Avicenne, Bobigny
  - HIA de Clermont-Tonnerre, Brest
  - CHU, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier Laennec, Creil
  - Centre Hospitalier Intercommunal, Créteil
  - Centre Hospitalier, Draguignan
  - Centre Hospitalier, Gap
  - Centre Hospitalier Robert Boulin, Libourne
  - Hôpital Le Cluzeau, Limoges
  - Centre Hospitalier Régional, Longjumeau
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - Centre Hospitalier F. QUESNAY, Mantes-la-Jolie
  - Institut Paoli Calmette, Marseille
  - Hôpital Nord APHM, Marseille
  - Centre Hospitalier Les Chanaux, Mâcon
  - Centre Hospitalier, Meaux
  - Centre Hospitalier Intercommunal, Meulan-en-Yvelines
  - Clinique du Pont de Chaume, Montauban
  - Centre Catalan d'Oncologie, Perpignan
  - Centre Hospitalier, Périgueux
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier de la Région d'Annecy (CHRA), Pringy
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper
  - Hôpital Pontchailloux, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Institut de Cancérologie de la Loire (I.C.L), Saint-Priest-en-Jarez
  - Centre Hospitalier de Salon de Provence, Salon-de-Provence
  - Centre Hospitalier, Sens
  - Centre Paul Strauss, Strasbourg
  - Hopital d'Instruction des Armées Sainte Anne, Toulon
  - Hôpital Larrey, Toulouse
  - Clinique Pasteur, Toulouse
  - Centre Hospitalier, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monnet I, Vergnenegre A, Robinet G, Berard H, Lamy R, Falchero L, Vieillot S, Schott R, Ricordel C, Chouabe S, Thomas P, Gervais R, Madroszyk A, Abdiche S, Chiappa AM, Greillier L, Decroisette C, Auliac JB, Chouaid C; GFPC 02-13 (METAL2) investigators. Phase III randomized study of carboplatin pemetrexed with or without bevacizumab with initial versus "at progression" cerebral radiotherapy in advanced non squamous non-small cell lung cancer with asymptomatic brain metastasis. Ther Adv Med Oncol. 2021 Apr 16;13:17588359211006983. doi: 10.1177/17588359211006983. eCollection 2021. PMID 33948123